CLINICAL TRIAL: NCT02956811
Title: DAPA-LVH - Does Dapagliflozin Regress Left Ventricular Hypertrophy In Patients With Type 2 Diabetes?
Brief Title: Does Dapagliflozin Regress Left Ventricular Hypertrophy In Patients With Type 2 Diabetes?
Acronym: DAPA-LVH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015DM07; 2016-000715-33 (EudraCT Number)
Record Dates: First submitted 2016-10-07; First posted 2016-11-07 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes; Left Ventricular Hypertrophy
Keywords: Type 2 Diabetes; Left Ventricular Hypertrophy; Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertrophy, Left Ventricular | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Dapagliflozin 10mg once daily for 12 months
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo 10mg once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — SGLT2 inhibitor
  Other Names: Forxiga
  Arms: Active
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Left ventricular hypertrophy (LVH) is common in people with type 2 diabetes (70%) and is the strongest independent risk factor for cardiovascular events and all-cause mortality that there is. It is worse than triple vessel coronary disease. LVH often occurs in patients with "normal" blood pressures (BP). Apart from BP, the other three main factors causing LVH are insulin resistance, obesity and cardiac preload. Dapagliflozin reduces ALL four factors known to promote LVH i.e. Dapagliflozin reduces weight, glycaemia, preload and blood pressure and is therefore the ideal agent to reduce LVH since it uniquely attacks all four known mediators of LVH. This trial will investigate the ability of dapagliflozin to regress LVH in 64 participants with normotensive diabetes. This will be done by seeing if dapagliflozin reduces left ventricular mass as measured by cardiac magnetic resonance imaging (MRI). This trial may identify a novel way to reduce the strong independent risk factor of LVH which often persists despite optimum medical therapy in patients with diabetes. If dapagliflozin does reduce LVH, this would be a key sign of which subgroup of patients with diabetes (those with LVH) should be especially targeted with dapagliflozin.

64 participants with type 2 diabetes and LVH will be recruited through the Scottish Diabetes Research Network (SDRN), Scottish Primary Care Research Network (SPCRN) and other routes, in this single centre study. Participants will be randomised to receive either 10mg dapagliflozin or placebo daily for 12 months. Cardiac MRI will be performed at baseline and at 12 months, this will be assessed for the primary outcome of change in left ventricular mass. Secondary outcomes will examine change in 24 hour blood pressure and weight.

DETAILED DESCRIPTION:
Left ventricular hypertrophy (LVH) is present in the majority of patients with type 2 diabetes, since it affects 70%. It is a strong independent predictor of cardiovascular deaths and events and is even worse than triple vessel coronary disease. The reason why LVH is so adverse is because it predates so many different cardiovascular events i.e. LVH is intrinsically arrhythmogenic and causes sudden death, it impedes left ventricular (LV) filling and leads to diastolic heart failure, it reduces coronary perfusion reserve and causes ischaemia and it causes left atrial enlargement, atrial fibrillation (AF), and cardio-embolic strokes. Controlling blood pressure (BP) and using a drug that blocks the renin-angiotensin system (RAS) are the standard approaches to the management of LVH but this approach is only partially effective since 44% of all patients with type 2 diabetes are normotensive patients with LVH. Thus "normotensive LVH" is very common. Indeed, BP only contributes 25% to the variability in LV mass seen in a population. (This is important since LVH is the same thing as a high level of LV mass). Despite a "normal" BP, normotensive LVH is just as risky as is hypertensive LVH. Nevertheless, we do know that regressing LVH irrespective of BP changes is an effective way to reduce the incidence of all major cardiovascular (CV) events including specifically sudden deaths, heart failure hospitalisations, new onset AF and strokes. The Losartan Intervention For Endpoint reduction in hypertension study (LIFE) provides conclusive proof that in diabetes, LVH regression per se reduces future cardiovascular events (by 24%), reduces CV deaths (by 37%) and reduces total deaths (by 41%) irrespective of BP.

Since controlling BP and using an angiotensin enzyme inhibitor or angiotensin receptor blocker is only partially effective at regressing LVH, additional ways of regressing LVH are now required. Insulin resistance is another mediator of LVH. The literature is awash with observational studies linking insulin resistance to LVH. Pub Med identifies 67 such papers, 5 of which are inconclusive. In the remaining 62 papers, 46 identify a significant relationship between LVH and some measure of insulin resistance while 16 found no such relationship. The large studies are mostly positive which includes Framingham, the Whitehall trial, the Strong Heart trial and the Women's Health Initiative trial while the Hypertension Genetic Epidemiology Network (HyperGEN) trial is the one large negative trial. There are a multitude of mechanisms whereby hyperinsulinaemia should produce LVH e.g. through signalling pathways such as Akt, transforming growth factor and peroxisome proliferator-activated receptors, through increased myocardial free fatty acid oxidation and through RAS activation causing sodium retention and thus increased cardiac preload. Therefore, it is likely that glycaemia contributes to LVH. However, reducing glycaemia per se appears to be insufficient to reduce CV events and key ancillary properties of each anti-glycaemic drug will be necessary to deliver the CV benefits we so badly need in diabetes.

A separate albeit related factor mediating LVH is obesity. Importantly, dapagliflozin has been shown to reduce weight. Thus the ideal treatment to regress LVH might be one that not only improves glycaemia but one that also aids weight loss. Dapagliflozin is the obvious option here since it has been shown to reduce both glycaemia and weight. Metformin is the only other anti-glycaemic which reduces both glycaemia and weight. Indeed the reason metformin reduces CV events in diabetes while other anti-glycaemic agents do not could well be in part because metformin reduces both glycaemia and weight which then reduce LVH (in fact we already have a separate British Heart Foundation grant to see if metformin really does reduce LV mass).

However dapagliflozin has other unique effects on the CV system which will impact on LVH. Dapagliflozin reduces blood pressure (LV afterload) and this by itself should also further reduce LVH. Further reducing BP even in normotensive patients has been shown to definitely regress LVH. Dapagliflozin also has diuretic effects which should reduce preload on the heart (this will be measured preload in this trial by MRI assessed end diastolic volume). The fact that dapagliflozin reduces both preload and afterload on the heart makes it uniquely promising as a way to reducing future CV events in patients with diabetes and, here, in reducing LV hypertrophy. Thus, dapagliflozin should regress LVH in patients with diabetes because it is unique in reducing the four main causes of LVH: glycaemia/insulin resistance, weight, preload and blood pressure. No other anti-diabetic medication alters even three of these. Even metformin only alters two since it does not change blood pressure. All other diabetic medications only reduce one (glycaemia) of these mediators of LVH. This may be why other new anti-glycaemic agents have failed to reduce CV events. In this trial, it is proposed to trial whether dapagliflozin causes regression of the independent cardiac risk factor of LVH in diabetic participants on optimal current evidence based therapy.

Original Hypothesis

Dapagliflozin will regress LVH in normotensive participants with type 2 diabetes.

RATIONALE FOR TRIAL

Cardiac MRI will be used to assess whether Dapagliflozin regresses LV mass more than placebo does over a one year treatment period. If it does, this would strongly suggest that Dapagliflozin will reduce CV events especially in the 44% of patients with type 2 diabetes who have LVH despite a controlled blood pressure.

All studies examining LVH regression require to be parallel group studies as effects on LV mass take 6-12 months to occur. Hence this is a parallel group, one year trial of the active drug vs. placebo.

The issue of what dapagliflozin does to CV events in diabetes is a hot topic. Most new antidiabetic drugs have been neutral or harmful but, judging by its pharmacological effects, it is quite possible that dapagliflozin might reduce CV events. A large ongoing trial (Dapagliflozin Effect on CardiovascuLAR Events - Thrombolysis in Myocardial Infarction (DECLARE - TIMI)) is just beginning to look at this. Why therefore do we also need to trial the effects of dapagliflozin on LV mass in those with LVH? If DECLARE-TIMI shows clearly that dapagliflozin reduces CV events, then our trial will have revealed a possible contributing mechanism to the reduced CV events i.e. LVH regression (patients in DECLARE-TIMI will not receive echocardiography so that subgroup analysis will not be able to answer this question and electrocardiograms are useless at identifying LVH. Furthermore, the accuracy of MRI over echo is so great that echo studies of LVH regression should no longer be considered reliable).

In other words, large mega-trials like DECLARE-TIMI are very valuable, but parallel smaller mechanistic studies like this can enhance their value by helping to explain the mechanisms producing the mega-trial results and/or helping to identify a subgroup who get a particular benefit meaning that the drug becomes more cost effective in that subgroup. Overall, this trial might, in conjunction with a mega-trial, help decide the course of future research (should LVH be a favoured target?) and help decide how to apply the results of a mega-trial in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent before any trial specific procedures.
2. Diagnosed with type 2 diabetes mellitus based on the current American Diabetes Association guidelines.
3. Aged >18 and <80 years
4. Body Mass Index ≥23
5. HbA1c 48-85mmol/mol (last known result within in the previous 6 months)
6. Blood pressure <145/90mmHg. Office BP at screening visit will be used however if this is above the inclusion criteria then the 24 hour or 16 hour recording at screening visit will be used to confirm that in the opinion of the PI the BP is adequately controlled.
7. Echocardiographic left ventricular (LV) hypertrophy (defined as an LV mass index of >115g/m2 for men and >95g/m2 for women indexed to body surface area or >48g/m2.7 or >44g/m2.7 when indexed to height) within the previous 6 months.
8. Women of childbearing potential must agree to take precautions to avoid pregnancy throughout the trial and for 4 weeks after intake of the last dose.

Exclusion Criteria:

1. 1. Any condition that in the opinion of the investigator may render the participant unable to complete the trial including non CV disease (e.g. active malignancy).
2. Participants with type 1 diabetes mellitus
3. Participants who have previously had an episode of diabetic ketoacidosis.
4. Serum Potassium or Sodium results outwith the normal range
5. Diagnosis of clinical heart failure
6. History of human immunodeficiency virus
7. LV systolic dysfunction (LVEF <45%) (last known result within in the previous 6 months)
8. eGFR <45ml/min (last known result within in the previous month)
9. Known liver function tests >3 times upper limit of normal (based on last measures and documented laboratory measurement in the previous 6 months)
10. Body weight >150Kg (unable to fit into a MRI scanner)
11. Contraindications to MRI (e.g. claustrophobia, metal implants, penetrative eye injury or exposure to metal fragments in eye requiring medical attention)
12. Past or current treatment with any SGLT2 inhibitor
13. Allergy to any SGLT2 inhibitor or lactose or galactose intolerance
14. Current treatment with loop diuretic
15. Currently receiving long term (>30 consecutive days) treatment with an oral steroid
16. Pregnant or breast feeding participants
17. Involvement in the planning and/or conduct of the trial (applies to Astra Zeneca or representative staff and/or staff at the trial site).
18. Participation in another interventional study (other than observational trials and registries) within 30 days before visit 1.
19. Individuals considered at risk for poor protocol or medication compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular (LV) Mass by Cardiac MRI at 52 weeks | Baseline and 52 weeks
  To see if Dapagliflozin reduces LV mass more than placebo in participants with type 2 diabetes and LV hypertrophy

SECONDARY OUTCOMES:
Change in 24 hour blood pressure (BP) recording at 52 weeks | Baseline and 52 weeks
  To confirm expected effect of dapagliflozin on BP
Change in Office blood pressure (BP) at 4, 17, 34 and 52 weeks | Baseline, 4, 17, 34 and 52 weeks
  To confirm expected effect of dapagliflozin on BP
Change in Body mass index at 4, 17, 34 and 52 weeks | Baseline 4, 17, 34 and 52 weeks
  To confirm expected effect of dapagliflozin on body mass index
Change in waist/hip ratio at 4, 17, 34 and 52 weeks | Baseline 4, 17, 34 and 52 weeks
  To confirm expected effect of dapagliflozin on waist/hip ratio
Change in waist circumference at 4, 17, 34 and 52 weeks | Baseline 4, 17, 34 and 52 weeks
  To confirm expected effect of dapagliflozin on waist circumference
Change in visceral fat massed with Abdominal MRI at 52 weeks | Baseline and 52 weeks
  To assess the effect of dapagliflozin on visceral fat mass.
Change in HbA1c at 4, 17, 34 and 52 weeks | Baseline, 4, 17, 34 and 52 weeks
  To assess the effects of dapagliflozin on HbA1c
Number of patients with adverse events related to treatment | 4, 17, 34 and 52 weeks
  Urinary symptoms and hypotensive symptoms will assess the tolerability of dapagliflozin in this patient group
Number of participants with abnormal laboratory values | 4, 17, 34 and 52 weeks
  Liver function tests will assess the tolerability of dapagliflozin in this patient group
Change in Fasting Insulin Resistance Index (FIRI) at 4, 17, 34 and 52 weeks | Baseline, 4, 17, 34 and 52 weeks
  To assess the effects of dapagliflozin on FIRI
Change in B-type Natriuretic Peptide (BNP) at 4, 17, 34 and 52 weeks | Baseline, 4, 17, 34 and 52 weeks
  To assess the effects of dapagliflozin on BNP
Change in uric acid at 4, 17, 34 and 52 weeks | Baseline, 4, 17, 34 and 52 weeks
  To assess the effects of dapagliflozin on uric acid
Change in diastolic function and global longitudinal strain | Baseline and 52 weeks
  To assess the effect of dapagliflozin on left ventricular diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MD, FRCP, Study Director — University of Dundee; Chim Lang, MD, FRCP, Principal Investigator — University of Dundee; Graeme Houston, FRCR, MBBCh, Study Director — University of Dundee; Rory McCrimmon, MBChB, MRCP, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dihoum A, Brown AJ, McCrimmon RJ, Lang CC, Mordi IR. Dapagliflozin, inflammation and left ventricular remodelling in patients with type 2 diabetes and left ventricular hypertrophy. BMC Cardiovasc Disord. 2024 Jul 12;24(1):356. doi: 10.1186/s12872-024-04022-7. PMID 38997620
- [Derived] Brown AJM, Gandy S, McCrimmon R, Houston JG, Struthers AD, Lang CC. A randomized controlled trial of dapagliflozin on left ventricular hypertrophy in people with type two diabetes: the DAPA-LVH trial. Eur Heart J. 2020 Sep 21;41(36):3421-3432. doi: 10.1093/eurheartj/ehaa419. PMID 32578850
- [Derived] Brown AJM, Lang C, McCrimmon R, Struthers A. Does dapagliflozin regress left ventricular hypertrophy in patients with type 2 diabetes? A prospective, double-blind, randomised, placebo-controlled study. BMC Cardiovasc Disord. 2017 Aug 23;17(1):229. doi: 10.1186/s12872-017-0663-6. PMID 28835229